CLINICAL TRIAL: NCT00033917
Title: Randomized Indomethacin Germinal Matrix Hemorrhage/Intraventricular Hemorrhage (GMH/IVH) Prevention Trial
Brief Title: Indomethacin Germinal Matrix Hemorrhage/Intraventricular Hemorrhage (GMH/IVH) Prevention Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Laura R. Ment, Professor Pediatrics and Neurology, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01NS027116 (NIH)
Record Dates: First submitted 2002-04-12; First posted 2002-04-15 (Estimated); Results first posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-02

CONDITIONS: Intraventricular Hemorrhage (IVH); Bleeding in the Brain; Prematurity; Very Low Birth Weight Infants
Keywords: intraventricular hemorrhage (IVH); bleeding in the brain; indomethacin; prematurity; very low birth weight infants
MeSH Terms: conditions — Premature Birth | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): indomethacin
  Interventions: Drug: indomethacin
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: indomethacin — an anti-inflammatory drug
  Arms: 1
Drug: placebo — saline
  Arms: 2

SUMMARY:
The purpose of this multicenter trial is to determine if indomethacin prevents bleeding in the brain of very low birth weight preterm infants.

DETAILED DESCRIPTION:
Intraventricular hemorrhage (IVH) or bleeding in the brain remains a major problem of preterm infants. This randomized, placebo-controlled multicenter trial enrolled 505 infants of 600 to 1250g birth weight to determine if indomethacin lowers the incidence of IVH, and 125 term infant controls. During this longitudinal trial, follow-up assessments have been performed at the ages of 3, 4 1/2, 6, 8, 12 and 16 years. The initial results at age 3 years revealed no advantages to the indomethacin group over and above the decreases in IVH, however, the results did show a significant increase in ventriculomegaly in the "placebo" group. Results at 4 1/2, 6 and 8 years of age showed beneficial effects of indomethacin on cognitive and behavioral outcomes over and above the effects on preventing IVH but not at later ages. At 12 and 16 years, no significant influence of indomethacin on cognitive outcome was noted.

Age, gender and zip-code matched control subjects were added when the preterm subjects were 8 years. Throughout all subsequent testing, term controls have higher IQ and Peabody Picture Vocabulary Scores.

Additional longitudinal volumetric, functional and diffusion tensor MR imaging studies showed differences between preterm and term control subjects at 8, 12 and 16 years of age. These were consistent with utilization of the right hemisphere and left cerebellum for language in the preterm group compared to term controls. No effects of indomethacin were seen.

The study closed on 31 March 2012.

ELIGIBILITY:
* Preterm infants < 1250 g birth weight
* Admitted to participating institution < 6 hrs of age
* No evidence for congenital malformations
* Cranial US at 6 postnatal hours without evidence of Grades III - IV intraventricular hemorrhage

Max Age: 6 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 630 (Actual)
Dates: Start 1989-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura R. Ment, M.D., Principal Investigator — Department of Pediatrics, Yale University School of Medicine
Locations (3):
- United States (3):
  - Yale University School of Medicine, New Haven, Connecticut
  - Maine Medical Center, Portland, Maine
  - Brown University School of Medicine, Providence, Rhode Island

REFERENCES:
- [Background] Ment LR, Oh W, Ehrenkranz RA, Philip AG, Vohr B, Allan W, Duncan CC, Scott DT, Taylor KJ, Katz KH, et al. Low-dose indomethacin and prevention of intraventricular hemorrhage: a multicenter randomized trial. Pediatrics. 1994 Apr;93(4):543-50. PMID 8134206
- [Background] Ment LR, Oh W, Ehrenkranz RA, Phillip AG, Vohr B, Allan W, Makuch RW, Taylor KJ, Schneider KC, Katz KH, et al. Low-dose indomethacin therapy and extension of intraventricular hemorrhage: a multicenter randomized trial. J Pediatr. 1994 Jun;124(6):951-5. doi: 10.1016/s0022-3476(05)83191-9. PMID 8201485
- [Background] Ment LR, Vohr B, Oh W, Scott DT, Allan WC, Westerveld M, Duncan CC, Ehrenkranz RA, Katz KH, Schneider KC, Makuch RW. Neurodevelopmental outcome at 36 months' corrected age of preterm infants in the Multicenter Indomethacin Intraventricular Hemorrhage Prevention Trial. Pediatrics. 1996 Oct;98(4 Pt 1):714-8. PMID 8885951
- [Background] Ment LR, Westerveld M, Makuch R, Vohr B, Allan WC. Cognitive outcome at 4 1/2 years of very low birth weight infants enrolled in the multicenter indomethacin intraventricular hemorrhage prevention trial. Pediatrics. 1998 Jul;102(1 Pt 1):159-60. doi: 10.1542/peds.102.1.159. No abstract available. PMID 9714645
- [Background] Ment LR, Vohr B, Allan W, Westerveld M, Sparrow SS, Schneider KC, Katz KH, Duncan CC, Makuch RW. Outcome of children in the indomethacin intraventricular hemorrhage prevention trial. Pediatrics. 2000 Mar;105(3 Pt 1):485-91. doi: 10.1542/peds.105.3.485. PMID 10699097
- [Background] Peterson BS, Vohr B, Staib LH, Cannistraci CJ, Dolberg A, Schneider KC, Katz KH, Westerveld M, Sparrow S, Anderson AW, Duncan CC, Makuch RW, Gore JC, Ment LR. Regional brain volume abnormalities and long-term cognitive outcome in preterm infants. JAMA. 2000 Oct 18;284(15):1939-47. doi: 10.1001/jama.284.15.1939. PMID 11035890
- [Background] Ment LR, Vohr B, Allan W, Katz KH, Schneider KC, Westerveld M, Duncan CC, Makuch RW. Change in cognitive function over time in very low-birth-weight infants. JAMA. 2003 Feb 12;289(6):705-11. doi: 10.1001/jama.289.6.705. PMID 12585948
- [Background] Ment LR, Peterson BS, Meltzer JA, Vohr B, Allan W, Katz KH, Lacadie C, Schneider KC, Duncan CC, Makuch RW, Constable RT. A functional magnetic resonance imaging study of the long-term influences of early indomethacin exposure on language processing in the brains of prematurely born children. Pediatrics. 2006 Sep;118(3):961-70. doi: 10.1542/peds.2005-2870. PMID 16950986
- [Background] Ment LR, Kesler S, Vohr B, Katz KH, Baumgartner H, Schneider KC, Delancy S, Silbereis J, Duncan CC, Constable RT, Makuch RW, Reiss AL. Longitudinal brain volume changes in preterm and term control subjects during late childhood and adolescence. Pediatrics. 2009 Feb;123(2):503-11. doi: 10.1542/peds.2008-0025. PMID 19171615
- [Background] Gozzo Y, Vohr B, Lacadie C, Hampson M, Katz KH, Maller-Kesselman J, Schneider KC, Peterson BS, Rajeevan N, Makuch RW, Constable RT, Ment LR. Alterations in neural connectivity in preterm children at school age. Neuroimage. 2009 Nov 1;48(2):458-63. doi: 10.1016/j.neuroimage.2009.06.046. Epub 2009 Jun 25. PMID 19560547
- [Background] Luu TM, Vohr BR, Schneider KC, Katz KH, Tucker R, Allan WC, Ment LR. Trajectories of receptive language development from 3 to 12 years of age for very preterm children. Pediatrics. 2009 Jul;124(1):333-41. doi: 10.1542/peds.2008-2587. PMID 19564317
- [Background] Myers EH, Hampson M, Vohr B, Lacadie C, Frost SJ, Pugh KR, Katz KH, Schneider KC, Makuch RW, Constable RT, Ment LR. Functional connectivity to a right hemisphere language center in prematurely born adolescents. Neuroimage. 2010 Jul 15;51(4):1445-52. doi: 10.1016/j.neuroimage.2010.03.049. Epub 2010 Mar 25. PMID 20347043
- [Background] Mullen KM, Vohr BR, Katz KH, Schneider KC, Lacadie C, Hampson M, Makuch RW, Reiss AL, Constable RT, Ment LR. Preterm birth results in alterations in neural connectivity at age 16 years. Neuroimage. 2011 Feb 14;54(4):2563-70. doi: 10.1016/j.neuroimage.2010.11.019. Epub 2010 Nov 10. PMID 21073965
- [Background] Luu TM, Vohr BR, Allan W, Schneider KC, Ment LR. Evidence for catch-up in cognition and receptive vocabulary among adolescents born very preterm. Pediatrics. 2011 Aug;128(2):313-22. doi: 10.1542/peds.2010-2655. Epub 2011 Jul 18. PMID 21768322
- [Background] Constable RT, Vohr BR, Scheinost D, Benjamin JR, Fulbright RK, Lacadie C, Schneider KC, Katz KH, Zhang H, Papademetris X, Ment LR. A left cerebellar pathway mediates language in prematurely-born young adults. Neuroimage. 2013 Jan 1;64:371-8. doi: 10.1016/j.neuroimage.2012.09.008. Epub 2012 Sep 12. PMID 22982585
- [Background] Reiss AL, Kesler SR, Vohr B, Duncan CC, Katz KH, Pajot S, Schneider KC, Makuch RW, Ment LR. Sex differences in cerebral volumes of 8-year-olds born preterm. J Pediatr. 2004 Aug;145(2):242-9. doi: 10.1016/j.jpeds.2004.04.031. PMID 15289777

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Preterm neonates of 600 - 1250 g birth weight were enrolled between 6 and 12 postnatal hours at Yale New Haven Hospital (New Haven, CT), Maine Medical Center (Portland, ME) and Women and Infants' Hospital (Providence, RI).
Pre-assignment Details: Cranial ultrasounds were performed on all study participants between 6 - 12 hours of age for group assignment. Subjects with major congenital cerebral malformations were excluded.
Groups:
- IVH Negative Indomethacin: Those subjects with no evidence for intraventricular hemorrhage (IVH) at 6 - 12 postnatal hours. These subjects were randomized to early low-dose indomethacin (0.1 mg/kg/d for 3 doses).
- IVH Negative Placebo: These subjects also had no evidence for IVH at 6 - 12 hours. They were randomized to an equal volume of placebo.
Period: Overall Study
Arm/Group | IVH Negative Indomethacin | IVH Negative Placebo
Started | 209 | 222
Completed | 209 | 222
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Indomethacin: subjects randomized to early low dose indomethacin
- Placebo: Group randomized to an equal volume of placebo
- Total: Total of all reporting groups
Arm/Group | Indomethacin | Placebo | Total
Number analyzed (Participants) | 209 | 222 | 431
Age Continuous [Mean (Standard Deviation); unit: hours] — Age is expressed in postnatal hours
  hours | 7.8 (2.3) | 7.9 (2.4) | 7.8 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 103 | 196
  Male | 116 | 119 | 235
Region of Enrollment [Number; unit: participants]
  United States | 209 | 222 | 431

OUTCOME MEASURES:

1. Primary Outcome: IVH at 5 Postnatal Days
Description: Cranial ultrasounds were performed daily for the first 5 postnatal days; the main outcome measure was intraaventricular hemorrhage (IVH) at 5 days of age
Time Frame: at 5 days
Population: All subjects had negative cranial ultrasounds with no evidence for IVH at 6 - 12 postnatal hours
Measure: Number; unit: IVH
Arm/Group | Indomethacin | Placebo
Number analyzed (Participants) | 209 | 222
IVH | 25 | 40

2. Secondary Outcome: Language Outcome
Description: Peabody Picture Vocabulary Test (PPVT) This is a semantic language test. The mean value is 100; standard deviation is 16 points. A higher score means better language; a lower score means poorer language.
  There are no subscales to the PPVT. The measurement unit is points on a scale. A score < 70 indicates severely abnormal language function.
Time Frame: at 8 years
Population: Three hundred twenty eight subjects were available at age 8 years. They were tested with the PPVT.
Measure: Number; unit: participants with PPVT score < 70
Groups:
- Indomethacin - no IVH: Subjects randomized to indomethacin and had no IVH
- Indomethacin - IVH: Randomized to indomethacin; had IVH
- Placebo - no IVH: Randomized to placebo - no IVH
- Placebo - IVH: Randomized to placebo; had IVH
Arm/Group | Indomethacin - no IVH | Indomethacin - IVH | Placebo - no IVH | Placebo - IVH
Number analyzed (Participants) | 145 | 20 | 135 | 28
participants with PPVT score < 70 | 12 | 5 | 24 | 7

ADVERSE EVENTS:
Time Frame: First 5 postnatal days
Arm/Group | IVH Negative Indomethacin | IVH Negative Placebo
Serious Adverse Events (participants affected / at risk) | 0/208 | 0/222
Other Adverse Events (participants affected / at risk) | 19/209 | 12/222
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVH Negative Indomethacin (N=209) | IVH Negative Placebo (N=222)
necrotizing enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) — x-ray diagnosis
decreased urine output (Renal and urinary disorders) | 19 (19) | 10 (10)
creatinine > 1.8 mg/dL (Renal and urinary disorders) | 5 (5) | 5 (5)
excessive bleeding (Blood and lymphatic system disorders) | 9 (9) | 10 (10)
platelets < 50,000 (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
ischemic changes by ECHO (Nervous system disorders) | 6 (6) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes